CLINICAL TRIAL: NCT00338845
Title: Safer Sex Intervention for At-risk Women in Mexico
Brief Title: Share Safer Sex Counseling Program for Changing Sexual Risk Behaviors in Mexican Female Sex Workers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas L. Patterson, Professor in Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH065849 (NIH); R01MH065849 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: STDs
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

ARMS (2):
- 1 (Experimental): Participants will receive the Share Safer Sex counseling program
  Interventions: Behavioral: Share Safer Sex program
- 2 (Active Comparator): Participants will receive a standard didactic safer-sex counseling session
  Interventions: Behavioral: Standard didactic safer-sex counseling program

INTERVENTIONS:
Behavioral: Share Safer Sex program — The Share Safer Sex intervention will consist of a single, 30 to 40 minute, one-on-one counseling session designed to increase personal awareness of the participant's current unsafe behaviors and the associated risks, help her understand her motivation to change, and increase her knowledge about how to practice safe sex. Demonstrations and practice exercises will be used to improve participants' attitudes about, as well as intentions to practice, condom use. The counseling session will include the following activities: assessing readiness for change; building motivation for change; and performing exercises in decisional balance, identification of problem and problem-solving, and knowledge and skill-building.
  Arms: 1
Behavioral: Standard didactic safer-sex counseling program — The standard counseling program will be based on a sexual risk reduction counseling program developed by the Centers for Disease Control and Prevention, and will focus on personal risk assessment and strategies for risk reduction. Additionally, it will incorporate risk reduction materials provided by CENSIDA, Mexico's National Center for AIDS Studies.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of the Share Safer Sex Program in reducing sexual risk behaviors among female sex workers in four Mexican cities close to the U.S. border.

DETAILED DESCRIPTION:
Mexican female sex workers (FSWs) represent a large portion of the reported cases of AIDS and other sexually transmitted diseases (STDs) in Mexico. Despite the imbalance in the distribution of reported cases, there have been few efforts to change high-risk sexual behaviors in this population. There has been a dramatic increase in HIV and other STDs over the past decade, especially in Mexican cities along the United States border. Border cities often have a thriving sex trade industry, and some are considered "sexual tourist" destinations. FSWs in these border cities, however, often do not know how to practice safe sex. A previous study showed that a culturally sensitive risk reduction counseling program was effective in reducing sexual risk behavior in FSWs in Tijuana, Mexico. It may therefore be possible to implement the same program, with similar efficacy, in other Mexican cities near the U.S. border. This study will evaluate the effectiveness of the Share Safer Sex Program versus a standard counseling program in reducing sexual risk behaviors among FSWs in the Mexican cities of Tijuana, Ciudad Juarez, Nuevo Laredo, and Matamoros.

Participants in this open label study will be randomly assigned to either the Share Safer Sex Program or a standard counseling program. Both programs will last for 6 months and will consist of a single counseling session lasting between 35 and 40 minutes. All participants will undergo blood collection and a gynecological exam upon study entry and 6 months later. The standard counseling program will be based on a sexual risk reduction counseling program developed by the Centers for Disease Control and Prevention, and will focus on personal risk assessment and strategies for risk reduction. Additionally, it will incorporate risk reduction materials provided by CENSIDA, Mexico's National Center for AIDS Studies. The Share Safer Sex Program will be tailored to the needs, values, beliefs, and behaviors of the participants, and will take into account gender and cultural differences. Counselors will work with participants to increase personal awareness of their current unsafe behaviors and the associated risks, help them understand their motivation to change, and increase their knowledge about how to practice safe sex. Demonstrations and practice exercises will be used to improve participants' attitudes about, as well as intentions to practice, condom use. The counseling session will include the following activities: assessing readiness for change; building motivation for change; and performing exercises in decisional balance, identification of problem and problem-solving, and knowledge and skill-building. Outcomes for both treatment groups will be assessed after 6 months. Participants in the standard counseling program will be offered an opportunity to participate in the Share Safer Sex Program upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Reports having had unprotected vaginal, oral, or anal sex at least once within 2 weeks prior to study entry

Exclusion Criteria:

* Consistent use of condoms or dental dams for vaginal, oral, and anal sex with all clients within 2 weeks prior to study entry
* Duration of employment as an FSW is less than 2 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2003-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected vaginal, oral, and anal sex with clients and spouse or steady partner | Measured at Month 6 post-treatment

SECONDARY OUTCOMES:
STD incidence | Measured at Month 6 post-treatment
Knowledge, self-efficacy, and positive outcome expectancies re: condom use | Measured at Month 6 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Patterson, PhD, Principal Investigator — Dept. of Psychiatry, University of California, San Diego
Locations (1):
- Study outreach clinic, Tijuana, B.c., Mexico

REFERENCES:
- [Result] Patterson TL, Mausbach B, Lozada R, Staines-Orozco H, Semple SJ, Fraga-Vallejo M, Orozovich P, Abramovitz D, de la Torre A, Amaro H, Martinez G, Magis-Rodriguez C, Strathdee SA. Efficacy of a brief behavioral intervention to promote condom use among female sex workers in Tijuana and Ciudad Juarez, Mexico. Am J Public Health. 2008 Nov;98(11):2051-7. doi: 10.2105/AJPH.2007.130096. Epub 2008 Sep 17. PMID 18799768
- [Result] Strathdee SA, Lozada R, Semple SJ, Orozovich P, Pu M, Staines-Orozco H, Fraga-Vallejo M, Amaro H, Delatorre A, Magis-Rodriguez C, Patterson TL. Characteristics of female sex workers with US clients in two Mexico-US border cities. Sex Transm Dis. 2008 Mar;35(3):263-8. doi: 10.1097/OLQ.0b013e31815b0. PMID 18032996
- [Result] Patterson TL, Semple SJ, Staines H, Lozada R, Orozovich P, Bucardo J, Philbin MM, Pu M, Fraga M, Amaro H, Torre Ade L, Martinez G, Magis-Rodriguez C, Strathdee SA. Prevalence and correlates of HIV infection among female sex workers in 2 Mexico-US border cities. J Infect Dis. 2008 Mar 1;197(5):728-32. doi: 10.1086/527379. PMID 18260766
- [Derived] Burgos JL, Gaebler JA, Strathdee SA, Lozada R, Staines H, Patterson TL. Cost-effectiveness of an intervention to reduce HIV/STI incidence and promote condom use among female sex workers in the Mexico-US border region. PLoS One. 2010 Jun 30;5(6):e11413. doi: 10.1371/journal.pone.0011413. PMID 20617193
- [Derived] Loza O, Patterson TL, Rusch M, Martinez GA, Lozada R, Staines-Orozco H, Magis-Rodriguez C, Strathdee SA; Proyecto Mujer Segura. Drug-related behaviors independently associated with syphilis infection among female sex workers in two Mexico-US border cities. Addiction. 2010 Aug;105(8):1448-56. doi: 10.1111/j.1360-0443.2010.02985.x. Epub 2010 Apr 27. PMID 20456292